CLINICAL TRIAL: NCT04347525
Title: The Effect of Culturally Adapted Cognitive Behaviour Therapy (CaCBT)-Based Guided Self Help in Depressed Patients With Myocardial Infarction. A Randomised Controlled Trial
Brief Title: The Effect of Culturally Adapted CBT-based Guided Self Help in Depressed Patients With Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peshawar Medical College (Other)
Collaborators: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Principal Investigator, Muhammad Irfan, Prof of Psychiatry & Director Research, Peshawar Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBT Post-MI LHR
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Infarction; Depression
Keywords: Cognitive Behaviour Therapy; Depression; Myocardial Infarction; Guided Self Help
MeSH Terms: conditions — Myocardial Infarction; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive CaCBT based guided self-help using the manual (Khushi Aur Khatoon) as an intervention in addition to treatment as usual
  Interventions: Other: CaCBT based guided self help using Khushi aur Khatoon Manual
- Control (No Intervention): This group will receive treatment as usual

INTERVENTIONS:
Other: CaCBT based guided self help using Khushi aur Khatoon Manual — CaCBT based guided self help using the manual named Khushi Aur Khatoon in the intervention arm
  Arms: Intervention

SUMMARY:
This is a randomized controlled assessor-blind clinical trial comparing CaCBT based guided self-help (using a manual titled Khushi Aur Khatoon) against treatment as usual (TAU)

DETAILED DESCRIPTION:
Among patients with heart disease, depression and anxiety disorders are extremely common. After a myocardial infarction (MI), depression tends to persist over the next year. Similarly, among individuals who have significantly elevated anxiety following an episode of acute coronary syndrome, only 50% have a resolution of their anxiety in the year after the event, which suggests that anxiety can remain a chronic problem for many patients. Depression confers a 2-fold increased risk of mortality and adverse cardiac events after MI or heart failure and has been linked to poor outcomes after cardiac surgery.

Cognitive behavioural therapy (CaCBT) is the best-studied form of psychotherapy in patients who have had a myocardial infarction, in reducing depressive symptoms. However, there is a dearth of literature on the use of psycho-social interventions in those with medical problems in low and middle-income countries. This study is planned to explore the effect of culturally adapted Cognitive Behavioural Therapy (CaCBT) based Guided self-help (using the book, Khushi Aur Khatoon) compared with treatment as usual in improving depression in MI patients. Participants visiting the Punjab Institute of Cardiology - Lahore, who meet the entry criteria will be randomly allocated to one of the groups, i.e., CaCBT (Intervention group) or TAU (Control Group) in a 1:1 ratio. after taking written informed consent.

With a 5% significance level and 90% power, it was calculated that 48 subjects per group were required for the trial, with a total number of 96. To accommodate up to 30% of the dropout, the participants plan to recruit 140 participants in the study.

Participants were assessed at baseline and 9-12 weeks (end of therapy) from baseline. The primary outcome measure was the Hospital Anxiety and Depression Scale (HADS). The secondary outcome measures include HADS Anxiety and Depression Subscales; Bradford Somatic Inventory (BSI) and World Health Organization Disability Assessment Schedule (WHO DAS 2.0). The participants also measured satisfaction with the treatment at the end of therapy using a visual analog scale.

The participants followed the CONSORT guidelines for reporting randomized controlled trials. The analyses were carried out on an intention-to-treat basis using SPSS version 25. Comparisons for intention-to-treat analysis participants were included in the groups to which they are randomized regardless of how long or even whether they received the treatment allocated to them or not. Missing values were imputed using the last observation carried forward (LOCF) method. Both Chi-Square and t-tests were used for baseline comparisons. End-of-therapy scores on various outcome measures between the Intervention and the Control groups were compared using an Analysis of Covariance (ANCOVA) to adjust for baseline scores.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Myocardial Infarction
* Score 8 or more on HADS
* Fulfilling criteria of Major Depressive Disorder using DSM-V

Exclusion Criteria:

* Participants with use of alcohol or drugs
* Significant cognitive impairment (intellectual disability or dementia)
* Active psychosis
* Participants who have received CBT during the previous 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale-Depression Subscale (HAD-D) | 9-12 weeks (end of therapy)
  Change in the score of the Hospital Anxiety and Depression Scale (HADS) from baseline to end of therapy. The total score is the sum of the 7 items, ranging from 0-21. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of depression.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A) | 9-12 weeks (end of therapy)
  Change in the score of the Hospital Anxiety and Depression Scale, Anxiety subscale (HADS-A) from baseline to end of therapy. The total score is the sum of the 7 items, ranging from 0-21. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety.
Bradford Somatic Inventory (BSI) | 9-12 weeks (end of therapy)
  Change in the score of Bradford Somatic Inventory (BSI) from baseline to end of therapy. Respondents rank each feeling item on a 5-point scale ranging from 0 (not at all) to 4 (extremely). Rankings characterize the intensity of distress during the past 7 days. Scores can be summed for each dimension, or calculated into each global index.
World Health Organisation Disability Assessment Schedule (WHODAS 2.0) | 9-12 weeks (end of therapy)
  Change in the score of World Health Organisation Disability Assessment Schedule (WHODAS 2.0) from baseline to end of therapy. The total score for WHODAS ranges from 0-100, where a high score indicates major living limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Farooq Naeem, PhD, Study Chair — University of Toronto
Locations (1):
- Punjab Institute of Cardiology, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No